CLINICAL TRIAL: NCT00161642
Title: A Phase 1 Dose Escalation Study of CMD-193 in Subjects With Advanced Malignant Tumors.
Brief Title: Study Evaluating CMD-193 in Advanced Malignant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3152K1-100
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2009-09-10 (Estimated); Status verified 2009-09

CONDITIONS: Neoplasms
Keywords: Malignant Tumors
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Drug: CMD-193

SUMMARY:
The purpose of this study is to determine the safety, tolerability and maximum tolerated dose of CMD-193. Preliminary information about how a person's body processes CMD-193 and how CMD-193 affects tumors will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant solid tumor that has progressed following standard therapy, or for which no standard effective treatment is available
* Tumor expression of Lewis Y antigen ( > or = 20% tumor cells positive for Lewis Y by immunohistochemistry assay)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Chemotherapy, radiation therapy, other cancer therapy, or investigational agents within 21 days of the first dose of CMD-193 (42 days if the previous chemotherapy included nitrosoureas or mitomycin C)
* Symptomatic or clinically active CNS metastases. Subjects who have had prior treatment with radiotherapy or surgical resection for CNS metastases will be permitted if CNS metastases have remained stable and have not required any treatment for at least 3 months prior to the first dose of CMD-193.
* Significant prior allergic reaction to recombinant human or murine proteins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2004-11; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Physical examinations
hematology panels
ECG

SECONDARY OUTCOMES:
Radiographic tumor evaluations
blood sampling for pharmacokinetic assessments

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (3):
- United States (3):
  - Lebanon, New Hampshire
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee